CLINICAL TRIAL: NCT07119957
Title: ProspEXPO : PROSPective Study of the Associations Between Hepatocellular Carcinoma and Chemical and Psychosocial Environmental EXPOsome
Brief Title: ProspEXPO : Study of the Associations Between Hepatocellular Carcinoma and Chemical and Psychosocial Environmental EXPOsome
Acronym: ProspEXPO
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 49RC25_0139; 2025-A00678-41 (Other: ANSM (French Health Ministry))
Record Dates: First submitted 2025-07-09; First posted 2025-08-13 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Cirrhoses, Liver; Carcinoma Liver
Keywords: Liver Cirrhosis; HepatoCellular Carcinoma (HCC); Exposome
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Cirrhosis | interventions — Blood Specimen Collection; Urination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): Group of patients with MASLD and/or ALD at cirrhosis stage, without HCC
  Interventions: Other: Blood, urine and stool biocollection
- Case group (Other): Group of patients with MASLD and/or ALD at cirrhosis stage and complicated by HCC
  Interventions: Other: Blood, urine and stool biocollection

INTERVENTIONS:
Other: Blood, urine and stool biocollection — Collection of blood, urine and stool sampling in order to build up a biocollection

SUMMARY:
The aim of the study is to build up a bio-collection of biological samples from patients with cirrhosis. Further work using this bio-collection will permit to describe the influence of different exposome factors (nutrition, physical activity, socio-demographic conditions, tobacco, alcohol, pollutants) on the occurrence of the main type of liver cancer (called HCC).

Indeed, in the vast majority of cases, HCC develops within cirrhosis, and the factors that precipitate the progression of cirrhotic patients to HCC remain largely unknown.

DETAILED DESCRIPTION:
It has recently emerged that various elements of the exposome (pollutants, societal and psycho-social determinants, addictions, etc.) influence and modulate individual HCC risk. Indeed, by interacting with conventional risk factors (alcohol, unbalanced diet, metabolic factors, smoking, genetic predisposition), environmental factors (such as chemicals, air pollution, occupational exposures) are thought to contribute to oxidative stress, inflammation and the hepatic immune response, leading to a tumorigenic milieu in the liver. Very recently, we demonstrated a relationship between a perfluoroalkyl compound and the severity of steatosis in MASLD. Societal and psycho-social determinants also influence liver disease and HCC risk via dietary "dysbiosis" and "addictive behaviours". A population-based study conducted in France by the FRANCIM network, looking at the influence of socio-economic environment and disparities on cancer survival in 19 major solid tumors, showed that disadvantaged areas were associated with poorer survival, including for HCC. Taken together, these findings demonstrate the need for further research into the links between HCC and exposure to toxic chemicals, lifestyle, and the social and psychosocial environment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of metabolic and/or alcoholic steatotic liver disease, as defined by the new nomenclature (MASLD, ALD, or mixed MetALD)
* Liver biopsy performed (less than 2 months ago) or planned as part of treatment for diagnosis of cirrhosis ("Control" group without HCC) or diagnosis of HCC on cirrhosis ("Case" group)
* Patient affiliated to or benefiting from a social security scheme
* Patient having signed an informed consent to participate in the study (bio-collection)

Exclusion Criteria:

* Causes of chronic liver disease other than MASLD, ALD, or MetALD
* Decompensation of cirrhosis in the two years prior to inclusion (ascites, hepatic encephalopathy, gastrointestinal variceal hemorrhage, liver failure, hepatorenal syndrome)
* For the "Control" group: history of hepatocellular carcinoma
* Pregnant, breast-feeding or parturient women
* Persons deprived of liberty by judicial or administrative decision

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Blood sample for biocollection | Baseline
  Blood samples will be collected in order to create a biocollection. Biological parameters will be defined only with future studies (no biological parameter scheduled for this study).
Urinary sample for biocollection | Baseline
  Urinary samples will be collected in order to create a biocollection. Biological parameters will be defined only with future studies (no biological parameter scheduled for this study).
faecal sample for biocollection | Baseline
  Faecal samples will be collected in order to create a biocollection. Biological parameters will be defined only with future studies (no biological parameter scheduled for this study).

CONTACTS AND LOCATIONS:
Overall Officials: Jérôme BOURSIER, Professor, Principal Investigator — Angers University Hospital
Locations (4):
- France (4):
  - Angers University Hospital, Angers
  - Centre Eugène Marquis (Oncology center), Rennes
  - Rennes University Hospital, Hepatogastroenteroly Department, Rennes
  - Tours University Hospital, HepatoGastroenterology Department, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kleiner DE, Brunt EM, Van Natta M, Behling C, Contos MJ, Cummings OW, Ferrell LD, Liu YC, Torbenson MS, Unalp-Arida A, Yeh M, McCullough AJ, Sanyal AJ; Nonalcoholic Steatohepatitis Clinical Research Network. Design and validation of a histological scoring system for nonalcoholic fatty liver disease. Hepatology. 2005 Jun;41(6):1313-21. doi: 10.1002/hep.20701. PMID 15915461
- [Background] Tron L, Remontet L, Fauvernier M, Rachet B, Belot A, Launay L, Merville O, Molinie F, Dejardin O, Francim Group, Launoy G. Is the Social Gradient in Net Survival Observed in France the Result of Inequalities in Cancer-Specific Mortality or Inequalities in General Mortality? Cancers (Basel). 2023 Jan 20;15(3):659. doi: 10.3390/cancers15030659. PMID 36765616
- [Background] Tron L, Belot A, Fauvernier M, Remontet L, Bossard N, Launay L, Bryere J, Monnereau A, Dejardin O, Launoy G; French Network of Cancer Registries (FRANCIM). Socioeconomic environment and disparities in cancer survival for 19 solid tumor sites: An analysis of the French Network of Cancer Registries (FRANCIM) data. Int J Cancer. 2019 Mar 15;144(6):1262-1274. doi: 10.1002/ijc.31951. Epub 2018 Dec 3. PMID 30367459
- [Background] David N, Antignac JP, Roux M, Marchand P, Michalak S, Oberti F, Fouchard I, Lannes A, Blanchet O, Cales P, Blanc EB, Boursier J, Canivet CM. Associations between perfluoroalkyl substances and the severity of non-alcoholic fatty liver disease. Environ Int. 2023 Oct;180:108235. doi: 10.1016/j.envint.2023.108235. Epub 2023 Sep 27. PMID 37776622
- [Background] Anstee QM, Reeves HL, Kotsiliti E, Govaere O, Heikenwalder M. From NASH to HCC: current concepts and future challenges. Nat Rev Gastroenterol Hepatol. 2019 Jul;16(7):411-428. doi: 10.1038/s41575-019-0145-7. PMID 31028350
- [Background] Singal AG, Llovet JM, Yarchoan M, Mehta N, Heimbach JK, Dawson LA, Jou JH, Kulik LM, Agopian VG, Marrero JA, Mendiratta-Lala M, Brown DB, Rilling WS, Goyal L, Wei AC, Taddei TH. AASLD Practice Guidance on prevention, diagnosis, and treatment of hepatocellular carcinoma. Hepatology. 2023 Dec 1;78(6):1922-1965. doi: 10.1097/HEP.0000000000000466. Epub 2023 May 22. No abstract available. PMID 37199193
- [Background] European Association for the Study of the Liver. EASL Clinical Practice Guidelines: Management of hepatocellular carcinoma. J Hepatol. 2018 Jul;69(1):182-236. doi: 10.1016/j.jhep.2018.03.019. Epub 2018 Apr 5. No abstract available. Erratum In: J Hepatol. 2019 Apr;70(4):817. doi: 10.1016/j.jhep.2019.01.020. PMID 29628281
- [Background] Huang DQ, Singal AG, Kono Y, Tan DJH, El-Serag HB, Loomba R. Changing global epidemiology of liver cancer from 2010 to 2019: NASH is the fastest growing cause of liver cancer. Cell Metab. 2022 Jul 5;34(7):969-977.e2. doi: 10.1016/j.cmet.2022.05.003. Epub 2022 Jun 3. PMID 35793659
- [Background] Niu X, Zhu L, Xu Y, Zhang M, Hao Y, Ma L, Li Y, Xing H. Global prevalence, incidence, and outcomes of alcohol related liver diseases: a systematic review and meta-analysis. BMC Public Health. 2023 May 11;23(1):859. doi: 10.1186/s12889-023-15749-x. PMID 37170239
- [Background] Younossi ZM, Golabi P, Paik JM, Henry A, Van Dongen C, Henry L. The global epidemiology of nonalcoholic fatty liver disease (NAFLD) and nonalcoholic steatohepatitis (NASH): a systematic review. Hepatology. 2023 Apr 1;77(4):1335-1347. doi: 10.1097/HEP.0000000000000004. Epub 2023 Jan 3. PMID 36626630
- [Background] Rinella ME, Lazarus JV, Ratziu V, Francque SM, Sanyal AJ, Kanwal F, Romero D, Abdelmalek MF, Anstee QM, Arab JP, Arrese M, Bataller R, Beuers U, Boursier J, Bugianesi E, Byrne CD, Castro Narro GE, Chowdhury A, Cortez-Pinto H, Cryer DR, Cusi K, El-Kassas M, Klein S, Eskridge W, Fan J, Gawrieh S, Guy CD, Harrison SA, Kim SU, Koot BG, Korenjak M, Kowdley KV, Lacaille F, Loomba R, Mitchell-Thain R, Morgan TR, Powell EE, Roden M, Romero-Gomez M, Silva M, Singh SP, Sookoian SC, Spearman CW, Tiniakos D, Valenti L, Vos MB, Wong VW, Xanthakos S, Yilmaz Y, Younossi Z, Hobbs A, Villota-Rivas M, Newsome PN; NAFLD Nomenclature consensus group. A multisociety Delphi consensus statement on new fatty liver disease nomenclature. J Hepatol. 2023 Dec;79(6):1542-1556. doi: 10.1016/j.jhep.2023.06.003. Epub 2023 Jun 24. PMID 37364790
- [Background] Goutte N, Sogni P, Bendersky N, Barbare JC, Falissard B, Farges O. Geographical variations in incidence, management and survival of hepatocellular carcinoma in a Western country. J Hepatol. 2017 Mar;66(3):537-544. doi: 10.1016/j.jhep.2016.10.015. Epub 2016 Oct 20. PMID 27773614
- [Background] Rumgay H, Arnold M, Ferlay J, Lesi O, Cabasag CJ, Vignat J, Laversanne M, McGlynn KA, Soerjomataram I. Global burden of primary liver cancer in 2020 and predictions to 2040. J Hepatol. 2022 Dec;77(6):1598-1606. doi: 10.1016/j.jhep.2022.08.021. Epub 2022 Oct 5. PMID 36208844